CLINICAL TRIAL: NCT00249483
Title: Placebo-Controlled Venlafaxine Treatment for Depressed Cocaine Abusers
Brief Title: Venlafaxine to Reduce Cocaine Dependence in Depressed Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #4706R NIDA-09236-14; P50DA009236 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine Addiction; Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Venlafaxine (Experimental): Venlafaxine 300mg daily
  Interventions: Drug: Venlafaxine

INTERVENTIONS:
Drug: Venlafaxine — Venlafaxiine 300mg/day
  Arms: Venlafaxine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Preliminary research has shown that venlafaxine, a medication currently used for treating depression, may also discourage cocaine use in depressed individuals. This study will evaluate the effectiveness of venlafaxine in reducing cocaine use and alleviating depression in individuals addicted to cocaine.

DETAILED DESCRIPTION:
Individuals addicted to cocaine often experience feelings of restlessness, irritability, and anxiety. They also often report feeling depressed when not using cocaine, and they tend to resume cocaine use to alleviate symptoms of depression. Venlafaxine is a medication that is currently used to treat depression and anxiety disorders. Preliminary research has shown that venlafaxine reduces depression, improves mood, and simultaneously reduces cocaine use in cocaine addicts. Further research is needed to confirm the benefits of venlafaxine for cocaine addicts. The purpose of this study is to evaluate the effectiveness of venlafaxine in reducing cocaine use, cocaine craving, and depression in individuals who are addicted to cocaine and diagnosed with depression.

This study will begin with a 1-week lead-in phase, during which all participants will receive placebo medication. Participants whose depression levels decrease will not continue in the treatment phase of the study, but will be eligible for cocaine relapse therapy and medication if deemed necessary by the treating psychiatrist. Participants who remain depressed following the lead-in phase will be randomly assigned to receive either venlafaxine or placebo for 12 weeks. Participants assigned to venlafaxine will initially receive a daily dose of 37.5 mg. After 4 days, the dose will be increased to 75 mg; each week thereafter, the dose will be increased by another 75 mg, up to a maximum of 300 mg per day, dependent on side effects and positive responses. Study visits will take place twice a week. At each visit, medication side effects and depression levels will be assessed, cocaine levels will be monitored with urine tests, and self-reports will be completed. Blood will be drawn once per month for laboratory tests. Participants will also attend a therapy session once a week, and they will meet with a psychiatrist every other week for assessments. Participants who show a decrease in depression during the 12 weeks of treatment will continue for an additional 12 weeks to further monitor cocaine use and depression levels.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV diagnosis criteria for current cocaine dependence
* Used cocaine at least one day in the month prior to study entry
* Meets DSM-IV criteria for major depression or dysthymia, with depression either primary (predates earliest life-time substance abuse), depression persistent during 6 months of cocaine abstinence in the past, or depression for at least 3 months prior to study entry
* If female, willing to use contraception throughout the study

Exclusion Criteria:

* Meets DSM-IV diagnosis criteria for bipolar disorder, schizophrenia, or any psychotic disorder other than transient psychosis due to drug abuse
* Chronic organic mental disorder
* Significant risk of suicide, based on current mental state or history
* Untreated seizure disorder or history of substance-related seizures
* Unstable physical disorders that may make study participation dangerous, including hypertension, hepatitis (mildly elevated transaminase levels that are less than 4 times the upper limit or normal levels are acceptable), and diabetes
* Coronary vascular disease, as indicated by medical history, suspected by abnormal ECG, or history of heart symptoms
* Irregular heartbeat as indicated by QRS duration greater than 0.11
* Current use of other prescribed psychotropic medications
* Currently meets DSM-IV diagnosis criteria for dependence on any drugs other than nicotine, marijuana, or alcohol
* History of allergic or adverse reaction to desipramine or venlafaxine
* Prior history of failing to respond to venlafaxine
* History of alcohol withdrawal syndrome in the year prior to study entry
* Current evidence of alcohol withdrawal, such as pulse rate greater than 115 beats per minute, blood pressure greater than 140/90 mm Hg, or visible tremors
* Pregnant or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 1999-10; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Cocaine use | baseline compared to 12 weeks of study or length of participation
  Proportion of patients achieving 3 weeks of cocaine abstinence based on self report and urine toxicology
Hamilton Depression Rating Scale | baseline compared to week 12 or last week of study participation
  Proportion of patients achieving a 50% reduction in HAM-D score at week 12 compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Kleber, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States